CLINICAL TRIAL: NCT03851757
Title: Cleansing Efficacy of Waist-shaped Interdental Brushes. A Randomized-controlled Crossover Study.
Brief Title: Cleansing Efficacy of Waist-shaped Interdental Brushes.
Acronym: Waist-shaped
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: AN5123
Record Dates: First submitted 2019-01-31; First posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-01

CONDITIONS: Periodontitis, Adult
Keywords: biofilm; interdental brushes; interproximal; oral hygiene; periodontal disease(s)/periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Intervention Model Description: Randomised, controlled, examiner-blinded, two-period crossover study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- waist-shaped interdental brush (Active Comparator): waist-shaped interdental brush, use four times per interdental space
  Interventions: Device: waist-shaped interdental brush
- cylindric interdental brush (Active Comparator): cylindric interdental brush, use four times per interdental space
  Interventions: Device: cylindric interdental brush

INTERVENTIONS:
Device: waist-shaped interdental brush — use four times each per interdental space
  Other Names: Brand name: Circum Topcaredent
  Arms: waist-shaped interdental brush
Device: cylindric interdental brush — use four times each per interdental space
  Other Names: Brand name: Topcaredent
  Arms: cylindric interdental brush

SUMMARY:
The aim of the present randomized and single-blinded cross-over study was to compare the cleansing efficacy of waist-shaped interdental brushes with that of cylindric interdental brushes in interproximal sites.

DETAILED DESCRIPTION:
Brushing efficacy of cylindric and waist-shaped interdental brushes was evaluated in a randomized, controlled, examiner-blinded, two-period crossover study. 20 periodontal maintenance patients of the University Hospital of Dental Prosthetics and Restorative Dentistry were recruited. Each subject was asked to attend three appointments. In the first visit (day one), baseline plaque and bleeding indices were assessed. Each proband was instructed by the same experienced dental hygienist with two sizes of waist-shaped and cylindric interdental brushes, respectively. Primary outcome measure plaque index and secondary outcome measure papillary bleeding index were assessed by two blinded and calibrated examiners at four sites per tooth.The odds ratio and confidence interval for establishing plaque free interdental sites were calculated with logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Periodontitis stage 3
* Completion of active periodontal treatment
* Maximum probing pocket depths of 5 mm
* No site ≥ 4 mm with bleeding on probing
* Bleeding on probing < 10%
* Open interproximal spaces both, in mandible and maxilla
* Presence of > 23 natural teeth with no need for prosthetic rehabilitation.

Exclusion Criteria:

* Oral or systemic diseases other than Periodontitis
* Mucosal / periodontal swelling or Suppuration
* Pregnancy
* Minority
* Need for frequent drug consumption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Turesky modification of the Quigley and Hein Plaque Index | 11 weeks
  This is a plaque index scored as 0 = no plaque; 1 = slight flecks of plaque at the cervical margin of the tooth; 2 = a thin continuous band of plaque (1 mm or smaller) at the cervical margin of the tooth; 3 = a band of plaque wider than 1 mm but covering < 1/3 of the crown of the tooth; 4 = plaque covering at least 1/3 but < 2/3 of the crown of the tooth or 5 = plaque covering 2/3 or more of the crown of the tooth. A higher grade is worse (more plaque) than a lower grade. After measuring plaque grades on four sites per tooh, the mode is calculated, which is defined as the plaque grade most often measured in an individual.

SECONDARY OUTCOMES:
papillary bleeding index by Saxer and Mühlemann | 11 weeks
  A periodontal probe is inserted into the gingival sulcus at the line angle on the mesial and distal aspect of the papilla and then moved coronally to the papilla tip (score 0 - no bleeding; score 1 - a single discreet bleeding point; score 2 - several isolated bleeding points or a single line of blood; score 3 - the interdental triangle fills with blood; score 4 - profuse bleeding occurs after probing and flows immediately into the marginal sulcus). A higher bleeding grade is worse (more inflammed tissues) than a lower grade. After measuring papillary bleeeding grades on four sites per tooh, the mode is calculated, which is defined as the papillary bleeding grade most often measured in an individual.

CONTACTS AND LOCATIONS:
Overall Officials: Ines Kapferer-Seebacher, Professor, Principal Investigator — Medical University of Innsbruck
Locations (1):
- Medical University of Innsbruck, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chongcharoen N, Lulic M, Lang NP. Effectiveness of different interdental brushes on cleaning the interproximal surfaces of teeth and implants: a randomized controlled, double-blind cross-over study. Clin Oral Implants Res. 2012 May;23(5):635-40. doi: 10.1111/j.1600-0501.2011.02387.x. Epub 2011 Dec 6. PMID 22146002
- [Background] Turesky S, Gilmore ND, Glickman I. Reduced plaque formation by the chloromethyl analogue of victamine C. J Periodontol. 1970 Jan;41(1):41-3. doi: 10.1902/jop.1970.41.41.41. No abstract available. PMID 5264376
- [Background] Saxer UP, Turconi B, Elsasser C. Patient motivation with the papillary bleeding index. J Prev Dent. 1977 Jul-Aug;4(4):20-2. No abstract available. PMID 351174
- [Derived] Schnabl D, Goebel G, Kadletz A, Gaenzer H, Steiner R, Laimer J, Kapferer-Seebacher I. Cleansing efficacy of waist-shaped inter-dental brushes. A randomized-controlled crossover study. J Clin Periodontol. 2020 Jan;47(1):30-35. doi: 10.1111/jcpe.13210. Epub 2019 Nov 3. PMID 31609489

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT03851757/Prot_SAP_000.pdf